CLINICAL TRIAL: NCT04369235
Title: Transcranial Electrical Stimulation With Special Waveform for Upper Extremity Rehabilitation for Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201702070
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-04

CONDITIONS: Stroke
Keywords: Stroke; Transcranial electrical stimulation; Upper-limb rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tCES & upper extremity rehabilitation (Experimental): The experiment group will receive tCES combined with upper extremity rehabilitation of affected side.
  Interventions: Device: tCES
- Sham tCES & upper extremity rehabilitation (Sham Comparator): The sham control group will receive sham tCES combined with upper extremity rehabilitation of affected side.
  Interventions: Device: Sham tCES

INTERVENTIONS:
Device: tCES — The positions of the lesion side primary motor cortex were defined as C3/C4 according to the international 10-20 system of electroencephalograms. tCES will be applied for 20 minutes at an intensity of 1.0 -1.5 mA direct current stimulation and a specific-added waveform each time, 3 times a week, lasting for 6 weeks.
  Arms: tCES & upper extremity rehabilitation
Device: Sham tCES — The positions of the lesion side primary motor cortex were defined as C3/C4 according to the international 10-20 system of electroencephalograms. Sham tCES will consist of a 5-second ramp up to 1.0-1.5 mA direct current stimulation and a specific-added waveform followed immediately by a 5-second ramp down, no current in the middle 19 minutes 40 seconds, and a ramp-up and ramp-down period during the last 10 seconds.
  Arms: Sham tCES & upper extremity rehabilitation

SUMMARY:
Transcranial electrical stimulation (tCES) is contemporarily important issues in the advanced rehabilitation medicine. tCES can selectively change the excitability of regional cortex with non-invansive and safety properties. Therefore, the investigators aim to develop a set of tCES system with special waveforms for using in clinical rehabilitation of upper extremities. This developed tCES system is smaller than all commercial available products, which could be conveniently and portably wore on head for clinical rehabilitation. In addition, the present tCES system with special waveforms developing by the investigators is much more efficient on improving neuroplasticity than the traditional transcranial direct current stimulation (tDCS) in rats. The investigators hope the tCES system combined with the rehabilitation of body extremities will become a routine treatment for stroke patients at hospitals or residential rehabilitation in the future.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) and intermittent theta burst stimulation (iTBS) were both demonstrated to have therapeutic potentials to rapidly induce neuroplastic effects in various rehabilitation training regimens. Recently, the investigators have developed a novel transcranial electrostimulation device that can flexibly output an electrical current with combined tDCS and iTBS waveforms. However, limited studies have determined the therapeutic effects of this special waveform combination on clinical rehabilitation. Herein, the investigators aiming to brain stimulation effects of tDCS-iTBS on upper-limb motor function in chronic stroke patients.

Twenty-four subjects with a chronic stroke were randomly assigned to a real non-invasive brain stimulation (NIBS; subjects received the real tDCS+iTBS output) group or a sham NIBS (subjects received sham tDCS+iTBS output) group. All subjects underwent 1 h treatment of a conventional rehabilitation program (3 days a week for 6 weeks), where a 20-min NIBS intervention was simultaneously applied during conventional rehabilitation. Outcome measures were assessed before and immediately after the intervention period: Fugl-Meyer Assessment-Upper Extremity (FMA-UE), Jebsen-Taylor Hand Function Test (JTT), and Finger-to-Nose Test (FNT).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 years.
2. Unilateral cerebral stroke with hemiplegia in Brunnstrom stage III-V.
3. 6 months to 5 years after stroke.
4. Adequate understanding of verbal/written information and physically able to complete the motor learning of functional tasks with the affected hand.

Exclusion Criteria:

1. Extremely sensitive to electrical stimulation and cannot tolerate it.
2. Contracture on upper extremities, and limitation in joint range of motion.
3. The muscle tone was severe spasticity.
4. Ossification or inflammation in muscle tissue.
5. A history of cardiopulmonary disease or arrhythmia.
6. With implantable medical electronic devices, like pacemaker.
7. Pressure sores or wounds on the skin of head and upper extremities.
8. Metal implants in the head (neck).
9. Severe cognitive or psychiatric disorders, such as schizophrenia or dissociative identity disorder.
10. A history of seizure or other brain pathology.
11. Brain surgery or severe brain trauma.
12. Drug or alcohol abuse.
13. Malignant neoplasm or rheumatism disorder, like SLE, RA, or AS.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Fugl-Meyer Assessment upper extremity scale (FMA-UE) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 6-week intervention (within 7 days after the last intervention session)
  The FMA-UE was performed (score ranges from 0 to 66) to assess upper limb motor recovery. Each movement is estimated by a 3-point scale (0-1-2). The total score of the FMA-UE is 66, and a higher score indicates that the patient has better movement ability.

SECONDARY OUTCOMES:
Change from baseline in the Jebsen-Taylor Hand Function Test (JTT) after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 6-week intervention (within 7 days after the last intervention session)
  The JTT assesses hand functions commonly used in activities of daily living. The subtests are scored according to time taken to complete the task. Total score is the sum of time taken for each subtest, with shorter times indicating better performance.
Change from baseline in the Finger to Nose Test after intervention | Baseline (within 7 days ahead to the 1st intervention session) and after 6-week intervention (within 7 days after the last intervention session)
  The Finger to Nose Test assesses coordination of upper-extremity movement. The number of complete nose-target movements during a 1 min period will be recorded.
Modified Ashworth scale (MAS) measures | Baseline (within 7 days ahead to the 1st intervention session) and after 6-week intervention (within 7 days after the last intervention session)
  The Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wei Peng, Ph.D., Principal Investigator — School of Biomedical Engineering, Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen SC, Yang LY, Adeel M, Lai CH, Peng CW. Transcranial electrostimulation with special waveforms enhances upper-limb motor function in patients with chronic stroke: a pilot randomized controlled trial. J Neuroeng Rehabil. 2021 Jun 30;18(1):106. doi: 10.1186/s12984-021-00901-8. PMID 34193179

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT04369235/Prot_SAP_000.pdf